CLINICAL TRIAL: NCT06540794
Title: Evaluation of the Respiratory Effects of Driving Pressure Guided Mechanical Ventilation Using Electrical Impedance Tomography in Patients Undergoing Robot-Assisted Laparoscopic Radical Prostatectomy
Brief Title: Evaluating Respiratory Effects of Driving Pressure Guided Mechanical Ventilation Using Electrical Impedance Tomography in Patients Undergoing Robot-Assisted Laparoscopic Radical Prostatectomy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ezgi Budak Ozyalcın, Medical Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 020724-982717
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-07

CONDITIONS: Prostate Cancer; Lung Protective Ventilation; Postoperative Pulmonary Complications
Keywords: driving pressure; electrical impedance tomography; robot assisted laparoscopic prostatectomy; peep titration; recruitment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group sPEEP (standard positive end-expiratory pressure) (No Intervention): Patients in this group will receive mechanical ventilation with a PEEP value of 5 cmH2O, following the recruitment maneuver.
- Group kPEEP (personalized positive end-expiratory pressure) (Experimental): A decremental PEEP titration strategy will be chosen after recruitment to determine the PEEP value that provides the lowest driving pressure. The personalized PEEP value (kPEEP) that provides the lowest driving pressure will be measured and maintained throughout the mechanical ventilation period. To find this value, the PEEP level will first be set at 15 cmH2O and maintained for 12 breathing cycles, after which the driving pressure will be recorded. Subsequently, the PEEP level will be decreased by 1 cmH2O and maintained for 12 breathing cycles, with the driving pressure recorded at each level. This strategy will continue until the PEEP level reaches 5 cmH2O. During these measurements, the tidal volume will be set at 8 ml/kg, the respiratory rate at 12 breaths/min, and the inspiratory: expiratory ratio at 1:2. The PEEP value that provides the lowest driving pressure will be recorded as kPEEP and maintained during pneumoperitoneum.
  Interventions: Other: PEEP TITRATION

INTERVENTIONS:
Other: PEEP TITRATION — Determining the optimal PEEP value that provides the lowest driving pressure using decremental PEEP titration.
  Arms: Group kPEEP (personalized positive end-expiratory pressure)

SUMMARY:
Robot-Assisted Laparoscopic Radical Prostatectomy is a method increasingly used for prostate cancer due to fewer complications, morbidity, and mortality compared to other methods. The technique involves inflating the abdomen with carbon dioxide to provide visualization and working in a steep Trendelenburg position, which puts pressure on the lungs and can cause them to collapse. The functional residual capacity reduction caused by general anesthesia, combined with the negative effects of the position, increases the risk of significant respiratory system complications during and after surgery.

Lung protective ventilation strategies can reduce the incidence of postoperative pulmonary complications (PPC) by alleviating iatrogenic injury to previously healthy lungs. Apart from a low tidal volume (VT), applying positive end-expiratory pressure (PEEP) can minimize the risk of atelectasis and/or overdistension.

There is limited information on how to adjust optimal PEEP under increased intra-abdominal pressure during laparoscopy. A meta-analysis study on acute respiratory distress syndrome (ARDS) patients showed that high driving pressure (plateau pressure - PEEP) is the most associated value with mortality. It was shown that VT, plateau pressure, and PEEP are not related to patient outcomes or only when they affect driving pressure. Subsequent retrospective and prospective studies confirmed the importance of driving pressure in ARDS patients and surgical patients.

For patients under mechanical ventilation, applying a personalized PEEP that provides the lowest driving pressure, along with maneuvers to open closed alveoli (recruitment), reduces respiratory system complications during and after surgery. One method to visualize the effects of these maneuvers and the ideal PEEP application, which provides the lowest driving pressure for the patient, is electrical impedance tomography (EIT), a non-invasive, radiation-free bedside imaging technique.

EIT, measured with 16 electrodes placed on an elastic belt around the patient's 4th to 6th ribs, shows impedance changes in the lungs. This method successfully visualizes and evaluates dynamic changes in gas distribution within the lungs and has been validated by computed tomography scans, proving safe for use in both adults and pediatric patients. EIT divides the lungs into four layers from ventral to dorsal, showing the percentage distribution of tidal volume in these regions. Examining the relative impedance changes allows for observing gas volume distribution entering the lungs and evaluating regional lung characteristics.

Therefore, EIT can contribute to examining the PEEP value that ensures homogeneous gas distribution in the lungs and preventing ventilator-associated lung injury.

The aim of our study is to evaluate the effect of driving pressure guided mechanical ventilation on lung gas distribution during robot-assisted laparoscopic radical prostatectomy through respiratory parameters recorded by EIT during surgery and perioperative period and to compare perioperative pulmonary complications with traditional ventilation methods

DETAILED DESCRIPTION:
General anesthesia increases the risk of respiratory complications and impairs arterial oxygenation by causing atelectasis in the dorsal regions of the lungs. Postoperative pulmonary complications (PPC) represent events such as atelectasis, pulmonary edema, pneumonia, pleuritis, reintubation, and the need for oxygen support after surgery, and are associated with increased morbidity, mortality, intensive care, and hospital stay durations, as well as higher healthcare costs. The effective strategy to reduce the incidence of PPC in patients under general anesthesia is still not clear.

Robot-assisted surgeries are increasingly preferred for prostatectomy, a curative treatment for prostate cancer, due to advantages such as less blood loss, less scar tissue formation, and shorter hospital stays compared to other surgical methods. During robotic surgery, many factors such as laparoscopy, pneumoperitoneum, and extreme Trendelenburg position can negatively affect lung function. Studies have shown that high driving pressure values, resulting from the set tidal volume target and PEEP values during mechanical ventilation, increase postoperative pulmonary complications.

Developing mechanical ventilation strategies based on personalized PEEP values that provide the lowest driving pressure after recruitment maneuvers to include closed alveoli in respiration and monitoring the effects of this method on the lungs during the perioperative period using electrical impedance tomography (EIT) is a highly useful tool. EIT, a non-invasive, radiation-free bedside monitoring system that detects real-time regional ventilation changes, can be used to guide individualized protective ventilation strategies to reduce perioperative respiratory system complications. Examining ROI values measured by EIT shows the effect of ventilation strategies on the distribution of tidal volume in the lungs. ROIs calculated by selecting layers, with ROI 1 and ROI 2 reflecting the ventral parts and ROI 3 and ROI 4 reflecting the dorsal parts, can be used to demonstrate the effect of the chosen ventilation strategy on lung gas distribution through intergroup comparison.

The age, gender, height, weight, body mass index, diagnosis, ASA score, preoperative hemoglobin level, additional systemic diseases, smoking history, prostate-specific antigen level, Gleason score, and prostate volume of the patients will be recorded. All patients will be monitored with electrocardiogram (ECG), peripheral oxygen saturation (SpO2), invasive arterial pressure (systolic arterial pressure, diastolic arterial pressure, and mean arterial pressure), and electrical impedance tomography. Patients will be prospectively randomized into two groups; group assignments will be determined using a closed-envelope technique.

All patients will be preoxygenated with 80% FiO2, followed by induction of anesthesia with 2 mcg/kg fentanyl, 2 mg/kg propofol, and 0.6 mg/kg rocuronium. After orotracheal intubation, patients will be placed on mechanical ventilation in volume control-autoflow mode with 8 ml/kg tidal volume, 2 L/min fresh gas flow, 0.4 inspired fractional oxygen (FiO2), an inspiratory: expiratory ratio of 1:2, and a respiratory rate to achieve normocapnia (partial carbon dioxide pressure PaCO2: 35-45 mmHg). Recruitment maneuvers will be applied to all patients.

During the recruitment maneuver: with an inspiratory: expiratory ratio of 1:1, a respiratory rate of 12 breaths/min, ventilation with a tidal volume of 8 ml/kg will be applied for 1 minute at a PEEP level of 5 cmH2O. This will be followed by ventilation with a tidal volume of 10 ml/kg for 1 minute at 10 cmH2O PEEP, and finally, ventilation with a tidal volume of 12 ml/kg for 1 minute at 15 cmH2O PEEP.The mechanical ventilation strategies for the patients will be planned according to their group.

For all patients, systolic arterial pressure, diastolic arterial pressure, mean arterial pressure, heart rate, and SpO2 values will be recorded before induction, after intubation, at 5-minute intervals for up to 60 minutes after pneumoperitoneum and Trendelenburg position, at 60 minutes after Trendelenburg position , at 75 minutes after Trendelenburg position , at 90 minutes after Trendelenburg position, at 120 minutes after Trendelenburg position, at 180 minutes after Trendelenburg position, at 240 minutes after Trendelenburg position, before extubation, 5 minutes after extubation , at 60 minutes postoperatively , at 24 hours postoperatively , and at 48 hours postoperatively . Additionally, while the patient is on mechanical ventilation, peak pressure, plateau pressure, PEEP, mean airway pressure (MPaw), compliance, and end-tidal carbon dioxide values will also be recorded.

Intermittent arterial blood gas analysis with invasive arterial monitoring is a routine practice in our daily practice. Arterial blood gas analysis will be performed preoperatively, immediately after intubation, at 15, 60, and 120 minutes after pneumoperitoneum and Trendelenburg position, immediately before extubation, and 5 minutes after extubation, with pH, partial oxygen pressure (pO2), partial carbon dioxide pressure (pCO2), oxygenation index (pO2/FiO2), bicarbonate, lactate, and hemoglobin values recorded.

Anesthesia duration, perioperative fluid volume, perioperative blood loss and urine output, operation duration, pneumoperitoneum duration, mechanical ventilation duration, and vasoactive agent use duration will be recorded.

In all patients, ROI values measured by electrical impedance tomography, which we use routinely in our daily practice, will be recorded before intubation, immediately after intubation, at 15, 60, and 120 minutes after pneumoperitoneum and Trendelenburg position, immediately before extubation in the supine position, and 5 minutes after extubation.

Postoperative pulmonary complications in patients will be monitored using SpO2, fever, cough, and sputum history, as well as prolonged intubation if present, and the duration of oxygen support and the development of additional pathology will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ASA score of I-II-III according to the American Society of Anesthesiologists (ASA) physical status classification system
* Surgery duration is expected to be longer than 2 hours

Exclusion Criteria:

* Patients who underwent surgery requiring mechanical ventilation for more than 1 hour within 2 weeks before the operation
* Patients with a body mass index over 35
* Patients with large bullae or pneumothorax, those currently receiving oxygen support, those with severe respiratory disease
* Patients with severe heart failure classified as NYHA class III-IV by the New York Heart Association (NYHA), those with a pacemaker or cardiac defibrillator implant
* Patients with progressive neuromuscular disease
* Patients who refused to participate in the study were excluded.

Max Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ROI and GI index | peroperative
  The ROI values measured by electrical impedance tomography for all patients were recorded before intubation, immediately after intubation, at the 15th, 60th, and 120th minutes of pneumoperitoneum and Trendelenburg position, before extubation in the supine position, and 5 minutes after extubation. The GI index values, calculated using mathematical software with the EIT values recorded on the computer, were recorded before intubation, immediately after intubation, before extubation in the supine position, and 5 minutes after extubation.

SECONDARY OUTCOMES:
POSTOPERATIVE PULMONARY COMPLICATIONS | up to 2 days following surgery
  Postoperative pulmonary complications in patients will be monitored using SpO2, fever, cough, and sputum history, as well as prolonged intubation if present, and the duration of oxygen support and the development of additional pathology will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi B Ozyalcın, Medical Doctor, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Cerrahpasa Faculty of Medicine Department of Anesthesiology and Reanimation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided